CLINICAL TRIAL: NCT03714386
Title: A Multicentre, Open-label, Prospective, Randomized Study to Explore the Morbimortality in Patients Dialyzed With the Theranova HDx in Comparison to On-Line - Hemodiafiltration (Study MoTHER HDx)
Brief Title: Study to Explore Morbimortality in Patients Dialyzed With the Theranova HDx in Comparison to On-Line-Hemodiafiltration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Senefro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MoTHER HDx
Record Dates: First submitted 2018-09-28; First posted 2018-10-22 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-04

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- expanded hemodialysis (HDx) (Experimental): HDx therapies must be implemented following current clinical practices guidelines and procedures at the hospital. No additional actions are required. General rules will be applied regarding dialysis prescription
  Interventions: Device: A medium cut-off dialyzer will be used for HDx.
- online hemodiafiltration (HDF-OL) (Active Comparator): OL-HDF therapies must be implemented following current clinical practices guidelines and procedures at the hospital. No additional actions are required. General rules will be applied regarding dialysis prescription
  Interventions: Device: A synthetic high-flux dialyzer will be used for OL-HDF.

INTERVENTIONS:
Device: A synthetic high-flux dialyzer will be used for OL-HDF. — A synthetic high-flux dialyzer used for OL-HDF must be implemented following current clinical practices guidelines and procedures at the hospital. No additional actions are required. General rules will be applied regarding dialysis prescription
  Arms: online hemodiafiltration (HDF-OL)
Device: A medium cut-off dialyzer will be used for HDx. — A medium cut-off dialyzer used for HDx must be implemented following current clinical practices guidelines and procedures at the hospital. No additional actions are required. General rules will be applied regarding dialysis prescription
  Arms: expanded hemodialysis (HDx)

SUMMARY:
study to evaluate the safety and efficacy of Expanded Hemodialysis (HDx) compared to hemodiafiltration (HDF) in patients with chronic kidney disease in Spain for up to 36 months.

Approximately 700 patients will be included.

DETAILED DESCRIPTION:
This is an open-label, prospective, 1:1 randomized, parallel-group, study to evaluate the safety and efficacy of Expanded Hemodialysis (HDx) compared to hemodiafiltration (HDF) in patients with chronic kidney disease in Spain for up to 36 months.

Stable incident hemodialysis patients from hemodialysis in-hospital units and related satellite centers in Spain.

ELIGIBILITY:
Inclusion Criteria:

* End stage Renal Disease (ESRD) patients
* Age> 18 years old
* HD therapy three times per week for 3 months at least and a maximum of 24 months.

Exclusion Criteria:

* No informed consent provided
* Synthetic membrane allergy
* Pregnant, breastfeeding, or planning to become pregnant
* Active systemic diseases: liver cirrhosis, malignancy prior to enrollment (except basal cell skin or similar) and / or immunosuppressive treatment in the 3 months before the recruitment.
* Scheduled for living-donor transplantation within the study period
* Patients with a significant residual renal function (defined as Urea clearance >2,5 ml/min.
* Currently participating in another interventional clinical study or has participated in another interventional clinical study in the last 3 months that may interfere with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — >18 years
Enrollment: 700 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular morbility | every 3 months
  Occurring during the first 36 months after recruitment (consequence of dialisys) cardiovascular sintomatology (stroke, Acute Coronary Syndrome, Peripheral Arterial Disease, Ischemic Colitis.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Perez Garcia, PhD, Principal Investigator — Hospital Universitario Infanta Leonor
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blankestijn PJ. Do Medium Cut-Off Dialyzers Offer Any Clinical Benefit or Should We Focus on Hemodiafiltration? J Am Soc Nephrol. 2025 Jun 27;36(8):1473-1475. doi: 10.1681/ASN.0000000777. No abstract available. PMID 40577061